CLINICAL TRIAL: NCT00131248
Title: Cross-over Trial of Medical Treatment for GERD in Preterm Infants
Brief Title: Medical Treatment for Gastroesophageal Reflux Disease (GERD) in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kathleen Kennedy, Professor - Pediatrics-Neonatology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GERD
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Metoclopramide; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Anti-reflux Medications, then Placebo (group 1) (Other): 3-day course of anti-reflux medications, followed by 7-day course placebo, followed by 4-day course anti-reflux medications.
  All study medication administered via nipple or orogastric (OG) tube. Metaclopramide (anti-reflux) given in 0.1mg/kg/dose q6hrs, 30min. prior to feedings. Ranitidine, 3mg/kg/dose, q12hrs. Saline placebo at same respective volumes.
  Interventions: Drug: Metaclopramide; Drug: Ranitidine; Drug: placebo
- Placebo, then Anti-reflux Medications (Other): 3-day course placebo, followed by 7-day course anti-reflux medication, followed by 4-day course placebo.
  All study medication administered via nipple or OG tube. Metaclopramide (anti-reflux) given in 0.1mg/kg/dose q6hrs, 30min. prior to feedings. Ranitidine, 3mg/kg/dose, q12hrs. Saline placebo at same respective volumes.
  Interventions: Drug: Metaclopramide; Drug: Ranitidine; Drug: placebo

INTERVENTIONS:
Drug: Metaclopramide
Drug: Ranitidine
Drug: placebo

SUMMARY:
Study Question: In premature infants with apnea and/or bradycardia attributed to gastroesophageal reflux disease (GERD), does treatment with medications (acid blockers and motility agents), compared to placebo, reduce the frequency of apnea and bradycardia?

Background: Many clinicians believe that apnea and bradycardia in preterm infants may be caused by gastroesophageal reflux (GER), however, studies have failed to demonstrate even a temporal association between episodes of GER and apnea. There have been no prospective randomized trials of treatment for GERD in preterm infants with apnea or other symptoms attributed to GER.

Methods: A randomized, cross-over study will be performed. This cross-over design will provide the patient's clinician with unbiased information about the patient's response to treatment. The clinician can use this information in deciding whether or not to continue treatment after the two-week study period.

DETAILED DESCRIPTION:
Study Question: In premature infants with apnea and/or bradycardia attributed to GERD, does treatment with H2 blockers and prokinetic agents, compared to placebo, reduce the frequency of apnea and bradycardia?

Background: The incidence of gastroesophageal reflux (GER) has been reported in as many as 50% of healthy term infants and 63% of preterm infants. Anecdotal observations of apnea and bradycardia clustered around feedings or with an episode of vomiting have suggested to clinicians that apnea and bradycardia in preterm infants may be caused by reflux, however, studies have failed to demonstrate even a temporal association between episodes of GER and apnea. One retrospective study concluded that anti-reflux medications did not reduce the frequency of apnea in premature infants. There have been no prospective randomized trials of treatment for GERD in preterm infants with apnea or other symptoms attributed to GER. Despite the lack of evidence supporting a causal relationship between GER and respiratory problems in preterm infants and the lack of data regarding the efficacy or safety of the treatments for GERD, many clinicians continue to believe that GER causes respiratory symptoms in preterm infants and these infants are commonly treated with medications for GERD.

Specific aims: To determine whether medications for GER are effective in reducing respiratory symptoms attributed to GER.

Methods: A randomized, controlled masked cross-over study will be performed. The cross-over design will prevent evaluation of long-term outcomes but will increase the power to evaluate short-term outcomes by using the patient as his/her own control. This cross-over design will also provide the patient's clinician with unbiased information about the patient's response to treatment. The clinician can use this information in deciding whether or not to continue treatment after the two-week study period. This approach for making therapeutic decisions in individual patients has been described as an "N of 1" trial.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants < 37 weeks gestation at birth; currently less than 44 weeks postmenstrual age.
* Not currently receiving mechanical ventilation
* Clinical diagnosis of GER and apnea/bradycardia suspected by the clinicians to be related to the GER. (Supporting diagnostic test information, such as upper gastrointestinal series [UGI] studies and pH probes will be recorded but not required for study enrollment.)
* Attending physician plan to begin anti-reflux medications
* Infants may be included in the study if they are on continuous positive airway pressure (CPAP) or methylxanthines for treatment of apnea only if the clinicians are willing to maintain the same regimen for the two-week duration of the study.
* Stable feeding regimen

Exclusion Criteria:

* History of congenital neurological defect
* Imminent discharge (within 2 weeks)
* Parent refusal

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2004-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Kennedy, MD, MPH, Principal Investigator — University of Texas
Locations (1):
- Memorial Hermann Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Wheatley E, Kennedy KA. Cross-over trial of treatment for bradycardia attributed to gastroesophageal reflux in preterm infants. J Pediatr. 2009 Oct;155(4):516-21. doi: 10.1016/j.jpeds.2009.03.044. Epub 2009 Jun 21. PMID 19540518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants = premature infants, <36 weeks gestation at birth, recruited from NICU at a hospital in Houston, Texas,USA, between 2004-2009
Groups:
- Medications, Placebo, Medications (Group 1): 3-day course of anti-reflux medications, followed by 7-day course placebo, followed by 4-day course anti-reflux medications.
  All study medication administered via nipple or OG tube. Metaclopramide (anti-reflux) given in 0.1mg/kg/dose q6hrs, 30min. prior to feedings. Ranitidine, 3mg/kg/dose, q12hrs. Saline placebo at same respective volumes.
- Placebo, Medications, Placebo (Group 2): received 3-day course placebo, followed by 7-day course anti-reflux medication, followed by 4-day course placebo.
  All study medication administered via nipple or OG tube. Metaclopramide (anti-reflux) given in 0.1mg/kg/dose q6hrs, 30min. prior to feedings. Ranitidine, 3mg/kg/dose, q12hrs. Saline placebo at same respective volumes.
Period: Intervention 1 (3-day Course)
Arm/Group | Medications, Placebo, Medications (Group 1) | Placebo, Medications, Placebo (Group 2)
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (24 Hour)
Arm/Group | Medications, Placebo, Medications (Group 1) | Placebo, Medications, Placebo (Group 2)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Intervention 2 (7-day Course)
Arm/Group | Medications, Placebo, Medications (Group 1) | Placebo, Medications, Placebo (Group 2)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Washout 2 (24 Hours)
Arm/Group | Medications, Placebo, Medications (Group 1) | Placebo, Medications, Placebo (Group 2)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Intervention 3 (4-day Course)
Arm/Group | Medications, Placebo, Medications (Group 1) | Placebo, Medications, Placebo (Group 2)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 18 participants initially enrolled; 1 withdrew, leaving 17 participants analyzed.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.1 (0.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Bradycardia Episodes/Day
Time Frame: 7 days
Population: 18 participants originally enrolled, 1 withdrew, leaving 17 participants analyzed.
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Medications | Placebo
Number analyzed (Participants) | 17 | 17
episodes per day | 4.6 (3.1) | 3.6 (2.7)

ADVERSE EVENTS:
Description: Safety population include only those who received study intervention.
Arm/Group | Medications | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes